CLINICAL TRIAL: NCT05945368
Title: A Prospective, Single-arm, Phase II Trial of Eribulin in Combination With Trastuzumab and Pertuzumab for Neoadjuvant Therapy HER2-Positive Early or Locally Advanced Breast Cancer
Brief Title: A Trial of Eribulin in Combination With HP Neoadjuvant Therapy in Patients With for HER2-Positive BC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Qiang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-138
Record Dates: First submitted 2023-05-28; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: Early or locally advanced breast cancer; HER 2-positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eribulin+Trastuzumab + Pertuzumab (Experimental): * Eribulin mesylate, 1.4 mg/m², days 1 and 8;
  * trastuzumab, 8 mg/kg loading dose in cycle 1 and 6 mg/kg thereafter on day 1;
  * pertuzumab with a loading dose of 840 mg in cycle 1 and 420 mg in subsequent cycles on day 1; 21 days in a cycle of 4 cycles
  Interventions: Drug: Eribulin mesylate injection、Pertuzumab、Trastuzumab

INTERVENTIONS:
Drug: Eribulin mesylate injection、Pertuzumab、Trastuzumab — * Eribulin mesylate, 1.4 mg /m², day 1 and day 8;
  * Trastuzumab, 8 mg/kg load dose in the first cycle and 6 mg/kg in each subsequent cycle on day 1;
  * Pertuzumab, 840 mg load dose in the first cycle and 420 mg in each subsequent cycle on day 1; There are four cycles in 21 days
  Other Names: Eribulin+HP

SUMMARY:
To evaluate the pathology complete response rate (pathology Complete Response, pCR) of eribulin combined with trastuzumab + pertuzumab in neoadjuvant therapy for HER-2 positive early or locally advanced breast cancer.

DETAILED DESCRIPTION:
Breast cancer with positive HER-2 is sensitive to chemotherapy and targeted therapy, and double-target regimen containing trastuzumab and pertuzumab is the preferred regimen no matter in neoadjuvant, adjuvant or advanced first-line stage. A series of clinical studies have established the strong position of trastuzumab + pertuzumab in the neoadjuvant therapy of HER2-positive breast cancer, but it is still unclear which chemotherapy drugs have the best efficacy when combined with them. Eribulin mesylate is a potent microtubule inhibitor. It is used as a single agent for the treatment of locally relapsed or metastatic breast cancer that has been treated with at least two chemotherapy regimens in the past, because of its good therapeutic effect and small toxic side effects The role of advanced breast cancer treatment is increasingly prominent. Therefore, the investigators plan to conduct clinical studies to evaluate the efficacy and safety of Eribulin combined with trastuzumab and pertuzumab in neoadjuvant therapy for HER-2 positive breast cancer, so as to provide better treatment options for neoadjuvant chemotherapy for HER-2 positive breast cancer. The investigators expect that Erribulin combined with trastuzumab and pertuzumab can achieve comparable results. If the pCR rate in this study reaches 40%, follow-up randomized controlled studies will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Newly treated female patients ≥18 years old and ≤75 years old;
* ECOG score 0-1;
* The pathology of breast cancer meets the following criteria:

Histologically confirmed invasive breast cancer; Tumor stage: Early or locally advanced breast cancer (T1c-T2 and cN1-cN3 or T3-T4/ cN0-cN3, M0)

* Pathologically confirmed HER2-positive breast cancer (definition: +++ or ++ immunohistochemical results with FISH nodes) Page 5 has 24 pages Page 6 has 24 pages Fruit is positive);
* Known hormone receptor status (ER and PgR);
* The functional level of major organs must meet the following requirements (no blood transfusion within 2 weeks prior to screening, no use of litterocyte, Platelet enhancer);

  * Blood routine: neutrophil (ANC) ≥1.5×109/L; Platelet count (PLT) ≥100×109/L; Red blood Protein (Hb) ≥90 g/L;
  * Blood biochemistry: total bilirubin (TBIL) ≤1.5× upper limit of normal value (ULN); Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) ≤1.5×ULN; Alkaline phosphatase (ALP) ≤2.5×ULN; urine Nitrogen (BUN) (or urea) and creatinine (Cr) ≤1.5×ULN;
* Cardiac ultrasound: left ventricular ejection fraction (LVEF) ≥55%;
* For female patients who are not menopausal or have not been surgically sterilized: arrive after the last dose during treatment and study therapy Within six months, agree to abstain from sex or use an effective contraceptive method.
* Participate in this study voluntarily, sign informed consent, have good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

* Stage IV breast cancer;
* Other specific types of breast cancer;
* Antitumor therapy or radiation therapy for any malignancy within the previous 5 years, excluding cured cervix Subcutaneous carcinoma, basal cell carcinoma or squamous cell carcinoma;
* Also receiving antitumor therapy in other clinical trials;
* Had major non-breast cancer related surgery within 4 weeks prior to randomization, or had not yet undergone such surgery Complete recovery in progress. 6. Serious cardiovascular and cerebrovascular diseases or discomfort, including but not limited to the following diseases:

  * History of heart failure or systolic dysfunction (LVEF < 50%)
  * High risk of uncontrolled arrhythmia
  * Angina pectoris, acute myocardial infarction
  * Valvular heart disease of clinical significance
  * Poor hypertension control (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
* Known allergic history of drug components of the program;
* A history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency conditions, Or have a history of organ transplantation;
* Pregnant and lactating women, fertile women with a positive baseline pregnancy test, or patients in Patients of childbearing age who were unwilling to use effective contraception throughout the trial period;
* The patient has a serious concomitant disease or other comorbiditis that would interfere with planned treatment, or is considered unwell by the investigator In conjunction with any other circumstances involved in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Pathology Complete Response | 24 to 28 weeks
  Pathology Complete Response (pCR) was evaluated in pathology complete response (pathology Complete Response) of Eribulin combined with trastuzumab and pertuzumab in neoadjuvant therapy for early or locally advanced breast cancer with positive HER-2.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | At baseline, 12 and 24 weeks
  evaluate the safety
Quality of Life（QoL) questionnaire | At baseline, 12 and 24 weeks
  evaluate the quality of life of patients with HER-2 positive early or locally advanced breast cancer treated with eribulin in combination with trastuzumab and partuzumab
Overall response rate (ORR) | from the first drug administration up to the first occurrence of progression or death (up to 24 months)
  The propotion of subjects with CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, Doc, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- LI YuDong, Guanzhou, Guangdong, China